CLINICAL TRIAL: NCT00257374
Title: Pedialyte or Gatorade for Viral Gastroenteritis in Adults: a Randomized, Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gatorade
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — gatorade

INTERVENTIONS:
Drug: Gatorade, Pedialyte and New Solution

SUMMARY:
Background: Pedialyte and Gatorade are advocated for the treatment of dehydration in viral gastroenteritis, but there is limited evidence to support their use.

Objective: To examine the efficacy, safety and palatability of Pedialyte, Gatorade, and a New Oral Rehydration Solution (NS).

Design: Randomized double blind. Setting: Inpatient, community hospital. Patients/Interventions: 75 consecutive adult patients (m/f=44/33) admitted with viral gastroenteritis were randomized to receive Gatorade, Pedialyte or NS for 48 hours. A yogurt/rice diet was allowed ad libitum.

Measurements: Stool and urine output, electrolytes, fluid intake, body weight, hematocrit and palatability of solutions.

Limitations: Smaller sample size and higher drop out (20%).

ELIGIBILITY:
Inclusion Criteria:

* Subjects were included if they had mild-to-moderate diarrhea, with mildly sunken eyes and a clinical assessment of dehydration of less than 5%, a serum sodium concentration between 130-150 mEq/L, adequate general health and nutrition, a BUN/creatinine ratio of >20 and with a normal pulse rate for age and degree of fever and adequate skin turgor

Exclusion Criteria:

* Patients were excluded if they had hyperthermia (>39.0º C), serum sodium >150 mEq/L or <130 mEq/L, white cell count >15,000, bloody diarrhea (dysentery), abnormal cardiovascular or renal function or an underlying metabolic or nutritional disorder and most importantly, if the clinical assessment of dehydration was >7% that suggested a need for intravenous fluids.

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Satish SC Rao, MD,PhD, FRCP(LON), Principal Investigator — University of Iowa
Locations (1):
- Dept. of Gastroenterology & Infectious Disease, Osmania Medical College, Hyderabad, India